CLINICAL TRIAL: NCT06799806
Title: The Impact of the Therapeutic Virtual Reality Headset on Patient Anxiety in the Waiting Room Before Flexible Bronchoscopy in Vigil
Acronym: REVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHM-2024/S15/04
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Bronchial Fibroscopy
Keywords: virtual reality headset; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: single-center, prospective, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- virtual reality (Experimental): virtual reality headset
  Interventions: Device: virtual reality device

INTERVENTIONS:
Device: virtual reality device — 20 minutes session with virtual reality device

SUMMARY:
Bronchial fibroscopy is a frequently used procedure in the management of pneumology patients, and can be a source of anxiety, particularly while waiting for the examination.

Investigator's professional experience has shown us that many patients are anxious in the waiting room before a flexible bronchoscopy in vigile.

A great deal of research has been carried out into the use of virtual reality to reduce anxiety and pain during care but shortly before bronchoscopy. The innovative aspect is to target the patient's waiting time for the examination. Waiting is a highly anxiety-provoking time, and nurses play a vital role in supporting patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with no age or gender restrictions, seen on an outpatient basis at Le Mans Hospital.
* In whom bronchial fibroscopy is indicated.
* Person affiliated with or benefiting from a social security .
* Free, informed and written consent signed by the participant and the investigator (no later than the day of inclusion and before any examination required by the research).
* Patient able and willing to answer questionnaires

Exclusion Criteria:

* Patient refusing to participate in research
* Patient who has already undergone bronchoscopy in vigil
* Patient premedicated for bronchial fibroscopy (anxiolytic, etc.)
* Patients with a history of epilepsy or psychiatric pathology
* Patient with vertigo
* Patient uncooperative, demented or unable to tolerate headgear.
* patient under guardianship or curatorship
* Patients suffering from blindness or deafness
* Patient with known significant intolerance to screens and/or virtual reality devices
* Pregnant, nursing or parturient women
* Unscheduled patients: emergencies, etc.
* Hospitalized patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Anxiety assessment | Immediately after intervention
  Anxiety assessment is measured using a Numerical Rating Scale (NRS) from 0 to 10, supplemented by a self-assessment questionnaire before and after using the Therapeutic Virtual Reality Headset.

SECONDARY OUTCOMES:
Assessment of bronchoscopy realisation and sample collection | Immediately after intervention
  Assessment of whether bronchoscopy has been performed correctly in the vigile state, aas well as any sampling required, using a questionnaire completed by the nurse present during vigile flexible bronchoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Christine PETIT, Principal Investigator — Centre Hospitalier le Mans
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No